CLINICAL TRIAL: NCT02667067
Title: Clinical Study Protocol for the Investigation Of The Simplify® Cervical Artificial Disc
Brief Title: Investigation of the Simplify® Cervical Artificial Disc
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G140154
Record Dates: First submitted 2015-10-08; First posted 2016-01-28 (Estimated); Results first posted 2022-06-06 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Cervical Degenerative Disc Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anterior cervical discectomy & fusion (ACDF) (Other)
  Interventions: Device: Anterior Cervical Discectomy & Fusion
- Simplify Disc (Experimental): Simplify Disc
  Interventions: Device: Simplify Disc

INTERVENTIONS:
Device: Simplify Disc — Simplify Disc at one level in the cervical spine.
  Arms: Simplify Disc
Device: Anterior Cervical Discectomy & Fusion — This study will utilize a non-concurrent historical control with subject-level data on a parallel group design. The historical control group will be formed from the randomized ACDF arm (N=133) of the recently completed Kineflex®|C Disc trial.
  Other Names: ACDF
  Arms: Anterior cervical discectomy & fusion (ACDF)

SUMMARY:
This study is intended to demonstrate that the Simplify® Disc is at least as safe and effective as conventional anterior cervical discectomy and fusion (ACDF) when used to treat one level between C3 to C7 for cervical degenerative disc disease (DDD) defined as intractable radiculopathy (arm pain and/or a neurological deficit) with or without neck pain or myelopathy due to a single-level abnormality localized to the level of the disc space in subjects who are unresponsive to conservative management.

DETAILED DESCRIPTION:
The objective of this clinical study is to evaluate the safety and effectiveness of the Simplify® Disc for treatment of DDD compared to conventional ACDF for reconstruction of the disc space at one level between C3 to C7 for DDD defined as intractable radiculopathy (arm pain and/or a neurological deficit) with or without neck pain or myelopathy due to a single-level abnormality localized to the level of the disc space that is unresponsive to conservative management.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 60 years of age;
* Have symptoms of cervical degenerative disc disease (DDD) at one cervical level from C3 to C7 defined as intractable radiculopathy (arm pain and /or a neurological deficit) with or without neck pain or myelopathy due to a single-level abnormality localized to the level of the disc space and radiographic evidence of at least one of the following;

  1. Spondylosis (defined by the presence of osteophytes or dark disc) on CT or MRI or;
  2. Disc height decreased by ≥ 1 mm when compared to adjacent levels on radiographic film, CT, or MRI or
  3. Disc herniation on CT or MRI;
* Have at least one of the following radiculopathy or myelopathy symptoms in neck and/or arm;

  1. Pain or paresthesias in a specific nerve root distribution from C3 to C7,
  2. Decreased muscle strength of at least one level on the 0-5 scale, or
  3. Abnormal sensation, including hyperesthesia or hypoesthesia.
* Have at least one of the following:

  1. At least six weeks of prior conservative treatment (e.g., physical therapy and/or use of anti-inflammatory medications and muscle relaxants at the manufacturer's recommended therapeutic dose);
  2. The presence of progressive symptoms (e.g., increasing numbness or tingling) or
  3. Signs of nerve root compression.
* Have a Neck Disability Index (NDI) greater than or equal to 40 on a scale of 100 (moderate disability);
* Be appropriate for treatment using an anterior surgical approach;
* Be likely to return for all follow-up visits and
* Be willing and able to provide Informed Consent for study participation.

Exclusion Criteria:

* Marked cervical instability on resting lateral or flexion/ extension X-ray (translation > 3 mm or > 11 degrees rotation to that of either adjacent non-treatment level);
* Non discogenic neck pain or non discogenic source of symptoms (e.g., tumor, rotator cuff injury, etc.);
* Radiographic confirmation of severe facet disease or facet degeneration;
* Bridging osteophytes;
* Less than 2 degrees of motion at index level;
* Prior surgery at the level to be treated, except laminotomy without accompanying facetectomy;
* Prior fusion at any cervical level;
* More than one neck surgery via anterior approach;
* Previous trauma to the C3-C7 levels resulting in compression or bursting;
* Documented presence of a free nuclear fragment at cervical levels other than the study level;
* Axial neck pain only (no radicular or myelopathy symptoms);
* Symptomatic DDD at more than one cervical level;
* Severe myelopathy (less than 3/5 muscle strength);
* Any paralysis;
* Recent history (within previous six months) of chemical or alcohol dependence;
* Active systemic infection;
* Infection at the site of surgery;
* Prior disc space infection or osteomyelitis in the cervical spine;
* Any terminal, systemic or autoimmune disease;
* Metabolic bone disease (e.g., osteoporosis/osteopenia , gout, osteomalacia, Paget's disease);
* Any disease, condition or surgery which might impair healing, such as;

  1. Diabetes mellitus requiring daily insulin management,
  2. Active malignancy,
  3. History of metastatic malignancy.
* Current or extended use (> 6 months) of any drug known to interfere with bone or soft tissue healing;
* Known PEEK, ceramic, titanium allergy;
* Arachnoiditis;
* Significant cervical anatomical deformity at the index level or clinically compromised cervical vertebral bodies at the index level due to current or past trauma (e.g., by radiographic appearance of fracture callus, malunion, or nonunion) or disease (e.g., ankylosing spondylitis, rheumatoid arthritis);
* Currently experiencing an episode of major mental illness (psychosis, major affective disorder, or schizophrenia), or manifesting physical symptoms without a diagnosable medical condition to account for the symptoms, which may indicate symptoms of psychological rather than physical origin;
* Pregnancy at time of enrollment, or planning to become pregnant, since this would contraindicate surgery ;
* Use of spinal stimulator at any cervical level prior to surgery;
* Currently a prisoner;
* Currently involved in spinal litigation which may influence the subjects reporting of symptoms or
* Participation in any other investigational drug, biologic or medical device study within the last 30 days prior to study surgery.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2021-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Malone, Study Director — NuVasive
Locations (16):
- United States (16):
  - La Jolla, California
  - Orange, California
  - Santa Monica, California
  - Thornton, Colorado
  - Sarasota, Florida
  - Evanston, Illinois
  - Carmel, Indiana
  - Paducah, Kentucky
  - Shreveport, Louisiana
  - Egg Harbor, New Jersey
  - Lockport, New York
  - Charlotte, North Carolina
  - Addison, Texas
  - Plano, Texas
  - Tyler, Texas
  - Reston, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited across 16 clinical sites in the United States
Pre-assignment Details: This is a non-randomized study. The 117 ACDF subjects are a historical control group. (Kineflex C Study; NCT#00374413)
Groups:
- Anterior Cervical Discectomy & Fusion (ACDF): Anterior Cervical Discectomy & Fusion: This study utilized a non-concurrent historical control with subject-level data on a parallel group design. The historical control group was formed from the randomized ACDF arm (N=133) of the recently completed Kineflex®|C Disc trial.
Period: Overall Study
Arm/Group | Anterior Cervical Discectomy & Fusion (ACDF) | Simplify Disc
Started | 117 | 150
Completed | 96 | 139
Not Completed | 21 | 11

BASELINE CHARACTERISTICS:
Population: One hundred sixty-six (166) subjects were enrolled in the Simplify® Cervical Artificial Disc population. Of these, 16 Simplify® Cervical Artificial Disc subjects were training subjects. The historical ACDF control population included 133 subjects. Of these, 117 control subjects were retained in the final PS designed sample
Groups:
- Total: Total of all reporting groups
Arm/Group | Anterior Cervical Discectomy & Fusion (ACDF) | Simplify Disc | Total
Number analyzed (Participants) | 117 | 150 | 267
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.1 (7.0) | 43.0 (8.9) | 43.5 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 91 | 159
  Male | 49 | 59 | 108
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 10 | 17
  White | 103 | 131 | 234
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 9 | 16
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 117 | 150 | 267

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite Clinical Success (CCS) of Simplify Disc
Description: Individual success for the Simplify® Disc subjects is defined as at least a 15 point improvement in Neck Disability Index (NDI) Score at 24 months compared with baseline, maintenance or improvement in neurologic status at 24 months compared with baseline, no device failures or revision, reoperation, removal and/or supplemental fixation within 24 months of index procedure; and the absence of major adverse events within 24 months.
  Individual success for the control ADCF device subjects is defined as at least a 15 point improvement in NDI Score at 24 months compared with baseline, maintenance or improvement in neurologic status at 24 months compared with baseline, no device failures or revision, reoperation, removal and/or supplemental fixation within 24 months; and the absence of major adverse events within 24 months.
  NDI scale is reported in a range from 0 - 100, with 0 consistent with best ability to function and 100 with worst ability to function.
Time Frame: Baseline, 24 Months
Population: Success is presented on observed data only
Measure: Count of Participants; unit: Participants
Arm/Group | Anterior cervical discectomy & fusion (ACDF) | Simplify Disc
Number analyzed (Participants) | 96 | 142
Participants | 68 | 132
Statistical Analysis 1: Comparison: Anterior cervical discectomy & fusion (ACDF) vs Simplify Disc; Test type: Superiority; p < .001, t-test, 1 sided

2. Secondary Outcome: Number of Subjects With 15-point Improvement in NDI at 3 Months (Time to Recovery)
Description: Time to recovery is defined as time to first 15-point improvement in NDI NDI scale is reported in a range from 0 - 100, with 0 consistent with best ability to function and 100 with worst ability to function.
Time Frame: Baseline, 3 Months
Population: Data is presented on available NDI scores.
Measure: Count of Participants; unit: Participants
Arm/Group | Anterior cervical discectomy & fusion (ACDF) | Simplify Disc
Number analyzed (Participants) | 111 | 145
Participants
  15-Point Improvement (Yes) | 90 | 139
  15-Point Improvement (No) | 21 | 6

3. Secondary Outcome: VAS Neck and Arm Pain
Description: Changes of at least 20 mm on a 100mm will be regarded as clinically significant VAS 0mm (no pain); VAS 100mm (worst pain)
Time Frame: Baseline, 24 Months
Population: Presented data available for comparison (preop and at month 24)
Measure: Count of Participants; unit: Participants
Arm/Group | Anterior cervical discectomy & fusion (ACDF) | Simplify Disc
Number analyzed (Participants) | 95 | 139
Participants
  Success | 83 | 134
  Failure | 12 | 5

4. Secondary Outcome: Neurological Status
Description: Neurological success was defined as maintenance or improvement in neurologic status at Month 24 as compared to baseline, as determined by the independent Clinical Events Committee (CEC). The CEC reviews neurological exams of motor, sensory, reflex, clumsiness, atrophy, cramping, spasms, numbness, dysphagia, dysphonia, and myelopathic gait to make an adjudication determination.
Time Frame: Baseline, 24 Months
Population: Subjects were analyzed based on available 24-month data.
Measure: Count of Participants; unit: Participants
Arm/Group | Anterior cervical discectomy & fusion (ACDF) | Simplify Disc
Number analyzed (Participants) | 95 | 139
Participants
  Improved | 52 | 111
  Maintained | 38 | 27
  Deteriorated | 5 | 1

5. Secondary Outcome: SF-12 Physical Component Score (PCS) Maintenance or Improvement
Description: The PCS is a sub-score of the SF-12. The SF-12 is a multipurpose short form survey with 12 questions all selected from the SF-36 Health Survey. The questions were combined, scored, and weighted to create two scores that provide glimpses into mental and physical functioning and overall health-related-quality of life. Higher scores indicate better outcomes. Scores range from 0-50.
  Data was not collected on SF-12 in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Time Frame: Baseline, 24 Months
Population: Subjects analyzed based on available data at month 24. Data was not collected on SF-12 in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc
Number analyzed (Participants) | 138
Participants
  Maintenance or Improvement | 129
  Absence of Maintenance or Improvement | 9

6. Secondary Outcome: SF-12 Mental Component Score (MCS) Maintenance or Improvement
Description: The MCS is a sub-score of the SF-12. The SF-12 is a multipurpose short form survey with 12 questions all selected from the SF-36 Health Survey. The questions were combined, scored, and weighted to create two scores that provide glimpses into mental and physical functioning and overall health-related-quality of life. Higher scores indicate better outcomes. Scores range from 0-50.
  Data was not collected on SF-12 in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Time Frame: Baseline, 24 Months
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc
Number analyzed (Participants) | 138
Participants
  Maintenance or Improvement | 105
  Absence of Maintenance or Improvement | 33

7. Secondary Outcome: Patient Questionnaires- Treatment Satisfaction Health Survey-
Description: Question 1 - "how does the subject rate satisfaction with the treated received" was compared between groups at Month 24. Answer options ranged from very dissatisfied to very satisfied.
Time Frame: 24 Months
Population: Presented data on available survey responses at Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | Anterior cervical discectomy & fusion (ACDF) | Simplify Disc
Number analyzed (Participants) | 96 | 138
Participants
  Very Satisfied | 67 | 122
  Satisfied | 20 | 12
  Somewhat Satisfied | 5 | 2
  Somewhat Dissatisfied | 3 | 2
  Dissatisfied | 1 | 0
  Very Dissatisfied | 0 | 0

8. Secondary Outcome: Odom's Criteria Results
Description: Results at 24 months for the investigational Simplify® Disc and at 24 months for the control ACDF will also be categorized by the physician according to Odom's Criteria.
Time Frame: 24 Months
Population: Data presented on subject's with Odom's Criteria result at Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | Anterior cervical discectomy & fusion (ACDF) | Simplify Disc
Number analyzed (Participants) | 95 | 139
Participants
  Excellent | 64 | 121
  Good | 18 | 12
  Fair | 8 | 5
  Poor | 5 | 1

9. Secondary Outcome: Dysphagia Handicap Index (DHI)
Description: Dysphagia Handicap Index (DHI scale) for the investigational Simplify® Disc at 24 months compared to baseline. A higher score is indicative of a less desirable outcome. It is scored 0-100.
  Data was not collected on DHI in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Time Frame: Baseline, 24 Months
Population: Data analyzed based on available 24-month DHI scores. Data was not collected on DHI in the historical ACDF control group. Only Simplify Disc subjects are reported. This was pre-specified in the study design.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Simplify Disc
Number analyzed (Participants) | 138
score on a scale | -2.3 (8.6)

10. Secondary Outcome: Average Disc Height (Index Level)
Description: Change in average disc height (index level) was compared to the baseline measurements and scored by an independent core lab (MMI). Average disc height is calculated as the simple average of the anterior and posterior disc heights.
Time Frame: Baseline, 24 Months
Population: Data presented on available images at Month 24
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Anterior cervical discectomy & fusion (ACDF) | Simplify Disc
Number analyzed (Participants) | 91 | 135
millimeters | 1.46 (1.24) | 0.93 (0.87)

11. Secondary Outcome: Average Disc Height (Above the Index Level)
Description: Change in average disc height (Above the index level) was compared to the baseline measurements and scored by an independent core lab (MMI). Average disc height is calculated as the simple average of the anterior and posterior disc heights.
Time Frame: Baseline, 24 Months
Population: Data presented on available images at Month 24
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Anterior cervical discectomy & fusion (ACDF) | Simplify Disc
Number analyzed (Participants) | 91 | 137
millimeters | -0.05 (0.40) | 0 (0.23)

12. Secondary Outcome: Average Disc Height (Below the Index Level)
Description: Change in average disc height (below the index level) was compared to the baseline measurements and scored by an independent core lab (MMI). Average disc height is calculated as the simple average of the anterior and posterior disc heights.
Time Frame: Baseline, 24 Months
Population: Data presented on available images at Month 24
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Anterior cervical discectomy & fusion (ACDF) | Simplify Disc
Number analyzed (Participants) | 59 | 106
millimeters | -0.07 (0.26) | -0.07 (0.31)

13. Secondary Outcome: Superior Adjacent Level Disc Degeneration
Description: Outcome reports the number and percentage of subjects with adjacent level disc degeneration (ALDD) above the index level.
Time Frame: Baseline, 24 Months
Population: Data presented on available images at Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | Anterior cervical discectomy & fusion (ACDF) | Simplify Disc
Number analyzed (Participants) | 95 | 139
Participants
  None | 15 | 87
  Mild | 22 | 26
  Moderate | 36 | 20
  Severe | 20 | 3
  Unable to assess | 2 | 3

14. Secondary Outcome: Inferior Adjacent Level Disc Degeneration
Description: Outcome reports the number and percentage of subjects with adjacent level disc degeneration (ALDD) below the index level.
Time Frame: Baseline, 24 Months
Population: Data presented on available images at Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | Anterior cervical discectomy & fusion (ACDF) | Simplify Disc
Number analyzed (Participants) | 95 | 139
Participants
  None | 14 | 95
  Mild | 15 | 15
  Moderate | 23 | 16
  Severe | 10 | 2
  Unable to assess | 33 | 11

15. Secondary Outcome: Device Migration
Description: Device migration assesses significant movement of the implant postoperatively
Time Frame: Baseline, 24 Months
Population: Data presented on available images at Month 24
Measure: Count of Participants; unit: Participants
Arm/Group | Anterior cervical discectomy & fusion (ACDF) | Simplify Disc
Number analyzed (Participants) | 95 | 139
Participants
  None | 90 | 137
  Anterior | 0 | 0
  Posterior | 0 | 0
  Left | 0 | 0
  Right | 0 | 0
  Unable to assess | 5 | 2

16. Secondary Outcome: Facet Deterioration
Description: Facet degeneration was assessed using MRI for the investigational Simplify Disc at 24 months compared to baseline.
  Facet degeneration was not assessed in the ACDF historical control group, as there is no 24 month MRI. This was pre-specified in the study design.
Time Frame: Baseline, 24 Months
Population: Data presented on available images at Month 24. Facet degeneration was not assessed in the ACDF historical control group, as there is no 24 month MRI. This was pre-specified in the study design.
Measure: Count of Participants; unit: Participants
Arm/Group | Simplify Disc
Number analyzed (Participants) | 139
Participants
  None | 80
  Mild | 42
  Moderate | 9
  Severe | 1
  Unable to Assess | 7

ADVERSE EVENTS:
Time Frame: Adverse events were collected continuously throughout study follow-up period. Results are reported through study day 790.
Groups:
- Anterior Cervical Discectomy & Fusion (ACDF): Anterior Cervical Discectomy & Fusion: This study utilized a non-concurrent historical control with subject-level data on a parallel group design. The historical control group will be formed from the randomized ACDF arm (N=133) of the recently completed Kineflex®|C Disc trial.
Arm/Group | Anterior Cervical Discectomy & Fusion (ACDF) | Simplify Disc
All-Cause Mortality (participants affected / at risk) | 0/117 | 0/150
Serious Adverse Events (participants affected / at risk) | 16/117 | 17/150
Other Adverse Events (participants affected / at risk) | 65/117 | 89/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anterior Cervical Discectomy & Fusion (ACDF) (N=117) | Simplify Disc (N=150)
Infections (all other infections - NOT at cervical surgical site) (Infections and infestations) | 1 (2) | 2 (2)
Pseduoarthrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Trauma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Headache (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Radiculopathy (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1)
Psychological Illness (Psychiatric disorders) | 1 (1) | 1 (1)
Pain (narcotic given) (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Adjacent Segment Degeneration (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (3)
Surgery at a location other than the spine (Surgical and medical procedures) | 0 (0) | 2 (5)
Gastrointestinal Complications (Gastrointestinal disorders) | 0 (0) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Inflammation Conditions (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Esophageal Perforation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infection; localized to cervical surgical site (Infections and infestations) | 0 (0) | 1 (1)
Ischemia (Cardiac disorders) | 0 (0) | 1 (1)
Deep wound infection; localized to cervical surgical site (Infections and infestations) | 0 (0) | 1 (1)
Implant Collapse or Subsidence (Product Issues) | 1 (1) | 0 (0)
Pain (No Narcotic Given) (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Other (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anterior Cervical Discectomy & Fusion (ACDF) (N=117) | Simplify Disc (N=150)
Spasm (Musculoskeletal and connective tissue disorders) | 5 (6) | 23 (24)
Trauma (Injury, poisoning and procedural complications) | 7 (8) | 12 (12)
Other (Injury, poisoning and procedural complications) | 6 (8) | 13 (15)
Dysphagia (Gastrointestinal disorders) | 3 (3) | 8 (9)
Infections (All other infections NOT at cervical surgical site) (Infections and infestations) | 5 (7) | 8 (12)
Inflammation (Musculoskeletal and connective tissue disorders) | 12 (14) | 16 (18)
Adjacent Segment Degeneration (Musculoskeletal and connective tissue disorders) | 8 (8) | 10 (11)
Radiculopathy (Nervous system disorders) | 21 (29) | 29 (35)
Pain (No narcotic given) (Musculoskeletal and connective tissue disorders) | 15 (18) | 14 (15)
Compressive Neuropathy (Nervous system disorders) | 9 (10) | 4 (4)
Headache (Nervous system disorders) | 12 (14) | 6 (8)
Pain (Narcotic given) (Musculoskeletal and connective tissue disorders) | 21 (29) | 11 (11)
GI Complications (Gastrointestinal disorders) | 0 (0) | 8 (9)

LIMITATIONS AND CAVEATS:
ACDF data is presented as a historical control fusion group from the Kineflex®|C Disc trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication results vary per investigator and per clinical trial agreement.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-01): https://cdn.clinicaltrials.gov/large-docs/67/NCT02667067/Prot_SAP_000.pdf